CLINICAL TRIAL: NCT06905522
Title: A Pan-Ultrashort Regimen for Drug-susceptible and Drug-resistant Pulmonary Tuberculosis: A Multi-Center Randomized Controlled Trial
Brief Title: A PAN-USR TB Multi-Center Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shenzhen Third People's Hospital (Other)
Collaborators: First Affiliated Hospital of Zhejiang University (Other); Beijing Chest Hospital of Capital Medical University (Unknown); Shenyang Tenth People's Hospital (Other); The Sixth People's Hospital of the Xinjiang Uygur Autonomous Region (Unknown); The Fourth Hospital of Inner Mongolia Autonomous Region (Unknown); Guizhou Aerospace Hospital (Unknown)
Responsible Party: Principal Investigator, Shuihua Lu, Professor, Shenzhen Third People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMART-C2405002
Record Dates: First submitted 2025-01-02; First posted 2025-04-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — bedaquiline; sitafloxacin; Linezolid; Pyrazinamide; Isoniazid; Protons; Rifampin; Ethambutol; Moxifloxacin; pretomanid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Drug-susceptible TB (A1) (Experimental): 2 months (9 weeks) BLSZ regimen: The treatment involves the use of bedaquiline (B), linezolid (L), sitafloxacin (S), and pyrazinamide (Z) throughout the entire process. At the end of 2 months (9 weeks) of treatment, if the sputum smear is still positive or if clinical symptoms have not improved, the treatment duration can be extended to 13 weeks. After the extended treatment period (3 months or 13 weeks), if the sputum smear remains positive or if clinical symptoms have not been relieved, the patient should be switched to the standard treatment regimen, and the subject should be withdrawn from the study.
  Interventions: Drug: Bedaquiline (B); Drug: Sitafloxacin (S); Drug: Linezolid (L); Drug: Pyrazinamide (Z)
- Drug-resistant TB (A2) (Experimental): 2 months (9 weeks) BLSZ regimen: The treatment involves the use of bedaquiline (B), linezolid (L), sitafloxacin (S), and pyrazinamide (Z) throughout the entire process. At the end of 2 months (9 weeks) of treatment, if the sputum smear is still positive or if clinical symptoms have not improved, the treatment duration can be extended to 13 weeks. After the extended treatment period (3 months or 13 weeks), if the sputum smear remains positive or if clinical symptoms have not been relieved, the patient should be switched to the standard treatment regimen, and the subject should be withdrawn from the study.
  Interventions: Drug: Bedaquiline (B); Drug: Sitafloxacin (S); Drug: Linezolid (L); Drug: Pyrazinamide (Z)
- Drug-susceptible TB (B) (Active Comparator): 2HRZE/4HR (26 weeks): Four drugs-isoniazid (H), rifampicin (R), pyrazinamide (Z), and ethambutol (E)-are used during the first 2 months of the intensive phase. This is followed by 4 months of consolidation treatment, during which only isoniazid and rifampicin are used.
  Interventions: Drug: Pyrazinamide (Z); Drug: Isoniazid (H); Drug: Rifampicin (R); Drug: Ethambutol (E)
- Drug-resistant TB (C) (Active Comparator): 6 months (26 weeks) of BPaLM: The treatment involves the use of bedaquiline (B), pretomanid (Pa), linezolid (L), and moxifloxacin (M) throughout the entire course. If the sputum culture remains positive at 4 months, or if clinical symptoms are not relieved by 6 months, or if chest CT results show worsening at 6 months, the treatment may be extended to 9 months. If the patient chooses to withdraw from the study at 6 months, they are allowed to do so.
  Interventions: Drug: Bedaquiline (B); Drug: Linezolid (L); Drug: Moxifloxacin (M); Drug: Pretomanid (Pa)

INTERVENTIONS:
Drug: Bedaquiline (B) — The initial dose of bedaquiline is 400 mg daily for 2 weeks, followed by 200 mg three times a week.
  Arms: Drug-resistant TB (A2); Drug-resistant TB (C); Drug-susceptible TB (A1)
Drug: Sitafloxacin (S) — 200mg once daily
  Arms: Drug-resistant TB (A2); Drug-susceptible TB (A1)
Drug: Linezolid (L) — 600mg once daily
  Arms: Drug-resistant TB (A2); Drug-resistant TB (C); Drug-susceptible TB (A1)
Drug: Pyrazinamide (Z) — 20-30 mg/kg/day; 1000 mg for patients weighing <50 kg, 1500 mg for patients weighing ≥50 kg but <75 kg, and 2000 mg for patients weighing ≥75 kg.
  Arms: Drug-resistant TB (A2); Drug-susceptible TB (A1); Drug-susceptible TB (B)
Drug: Isoniazid (H) — 4-6 mg/kg once daily, 300 mg once daily
  Arms: Drug-susceptible TB (B)
Drug: Rifampicin (R) — 8-12 mg/kg once daily, 450 mg for patients weighing <50 kg, 600 mg for patients weighing ≥50 kg but <75 kg, and 750 mg for patients weighing ≥75 kg.
  Arms: Drug-susceptible TB (B)
Drug: Ethambutol (E) — 15-25 mg/kg once daily, 750 mg once daily
  Arms: Drug-susceptible TB (B)
Drug: Moxifloxacin (M) — 400mg once daily
  Arms: Drug-resistant TB (C)
Drug: Pretomanid (Pa) — 200mg once daily
  Arms: Drug-resistant TB (C)

SUMMARY:
Tuberculosis (TB) remains a major public health issue and one of the top ten causes of death from a single infectious disease worldwide. China is among the countries with the highest TB burden, ranking third globally for total TB cases and second for drug-resistant TB cases. PAN-TB is an innovative concept in TB treatment, aiming to develop a universal regimen effective for all forms of active TB, including both drug-susceptible and drug-resistant strains. The primary goal of the PAN-TB regimen is to simplify the treatment process, reduce costs, and improve treatment success rates. The ideal Target Regimen Profile (TRP) for PAN-TB includes superior efficacy compared to standard treatment for non-drug-resistant TB, a reduced treatment duration from the current 4-6 months to 2-3 months, and improved safety and tolerability. This project aims to explore a new ultra-short-course treatment regimen for both drug-sensitive (DS-TB) and drug-resistant TB (MDR/RR-TB), which aligns with the latest trends in TB treatment both domestically and internationally. The regimen also has significant practical implications for enhancing treatment efficacy and reducing patient burden. Furthermore, the study will explore the identification of new biomarkers closely linked to treatment outcomes over the course of full-cycle therapy.

ELIGIBILITY:
Inclusion criteria:

1. Age range from 18 to 65 years old, regardless of gender;
2. Clinical symptoms and/or pulmonary imaging (chest X-ray or chest CT) support the diagnosis of active pulmonary tuberculosis;
3. Microbiological testing (molecular or phenotypic) confirms the presence of Mycobacterium tuberculosis, whether resistant to rifampicin or not; Recommend using respiratory specimens for GeneXpert MTB/RIF testing;
4. Voluntarily sign the informed consent form for participating in this project and be able and willing to accept follow-up visits;
5. Willing to undergo HIV testing;
6. Willing to preserve samples including DNA;
7. For women with fertility, they have a negative serum or urine pregnancy test within 3 days before enroll the study and be willing to use effective contraceptive measures during the study period. Female subjects without fertility must have records of menopause, hysterectomy, bilateral oophorectomy, or bilateral tubal ligation. Acceptable forms of contraception include condoms, intrauterine devices, cervical caps with spermicides, and diaphragm with spermicides.

Exclusion criteria:

1. Prior to this study, patients who were diagnosed with active pulmonary tuberculosis and had received anti-tuberculosis treatment (including first-line and second-line anti-tuberculosis drugs);
2. Intolerance or allergy to any investigational drug (i.e., bedaquiline, linezolid, fluoroquinolones [including moxifloxacin, sitagliptin], pyrazinamide);
3. Resistance to any investigational drug (i.e., bedaquiline, linezolid, fluoroquinolones [including moxifloxacin, sitagliptin], pyrazinamide). The following detection methods can be used: tNGS or other drug sensitivity testing methods (such as GeneXpert MTB/XDR, dissolution curve method, phenotypic drug sensitivity, etc.);
4. Suffering from hematogenous disseminated tuberculosis or coexisting with extrapulmonary tuberculosis (as specified in this study, the scope of pulmonary tuberculosis includes: simple pulmonary tuberculosis, pulmonary tuberculosis + tuberculous pleurisy/bronchial tuberculosis/mediastinal lymph node tuberculosis. Extrapulmonary tuberculosis refers to tuberculosis other than the chest-related types mentioned above);
5. Presence of non-tuberculous mycobacteria or other microbial lung infections that affect treatment outcomes;
6. Simultaneously using drugs that affect the efficacy of this study or have contraindications for combination therapy;
7. Use of any immunosuppressive medication or systemic glucocorticoids for more than 2 weeks before screening;
8. Any medication currently used or planned to be used that is known to significantly prolong the QTc interval, including but not limited to: amiodarone, amitriptyline, chloroquine, chlorpromazine, cisapride, dipyridamole, itraconazole, procaine, quinidine, or sotalol;
9. Uncontrolled blood sugar in diabetes, with no likelihood of improving blood sugar status according to the judgment of the researchers;
10. HIV positive;
11. Coexisting with severe autoimmune diseases, severe liver and kidney dysfunction, psychiatric disorders, hematological disorders, or malignant tumors;
12. Laboratory parameters within 14 days prior to recruitment: (1) Serum AST and ALT levels ≥ 3 times the upper limit of normal (ULN); (2) Blood creatinine ≥ 2 times ULN; (3) Hemoglobin ≤ 70 g/L; (4) Platelet count ≤ 50 × 10^9/L; (5) Blood potassium levels are ≥ 5.5 mmol/L or ≤ 3.5 mmol/L;
13. ECG QTcF ≥450 ms (allowing for one re-test during the screening phase to reassess eligibility for inclusion); Presence of one or more risk factors that could cause QT interval prolongation, such as arrhythmia, myocardial ischemia, etc.; history or family history of long QT syndrome;
14. Women who are pregnant or breastfeeding;
15. Weight <30 kg, or ≥90 kg;
16. The patient has participated in clinical trials of other drugs within the past 3 months during the screening period;
17. Other conditions deemed unsuitable for participation in the study by the research doctors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Estimated)
Dates: Start 2025-06-18 (Actual); Primary Completion 2029-01 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Unfavorable outcomes | 12 months (52 weeks)
  Percentage of patients with unfavorable outcomes (failure, treatment interruption, death, loss to follow-up, re-treatment, recurrence) at 12 months (52 weeks) after randomization
Safety | 2 months (9 weeks)
  Percentage of patients who have treatment interruption due to any reason or died within 2 months (9 weeks) after randomization

SECONDARY OUTCOMES:
Sputum culture conversion rate | 2 months (9 weeks) after randomization
Unfavorable outcomes (short-term) | 6 months (26 weeks) after randomization
Unfavorable outcomes (mid-term) | 18 months (78 weeks) after randomization
Time to sputum culture conversion | Median time
Serious adverse events or grade 3 or higher adverse events (short-term) | 12 months (52 weeks) after randomization
Serious adverse events or grade 3 or higher adverse events (mid-term) | 18 months (78 weeks) after randomization
Adverse events during treatment | 9 or 13 weeks (A1, A2); 26 weeks (B, C)
QTcF prolongation during treatment | 9 or 13 weeks (A1, A2); 26 weeks (B, C)
Liver function damage during treatment | 9 or 13 weeks (A1, A2); 26 weeks (B, C)

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Chest Hospital of Capital Medical University, Beijing
  - Shenzhen Third People's Hospital, Shenzhen
  - The Sixth People's Hospital of the Xinjiang Uygur Autonomous Region, Ürümqi

REFERENCES:
- [Result] Paton NI, Cousins C, Suresh C, Burhan E, Chew KL, Dalay VB, Lu Q, Kusmiati T, Balanag VM, Lee SL, Ruslami R, Pokharkar Y, Djaharuddin I, Sugiri JJR, Veto RS, Sekaggya-Wiltshire C, Avihingsanon A, Sarin R, Papineni P, Nunn AJ, Crook AM; TRUNCATE-TB Trial Team. Treatment Strategy for Rifampin-Susceptible Tuberculosis. N Engl J Med. 2023 Mar 9;388(10):873-887. doi: 10.1056/NEJMoa2212537. Epub 2023 Feb 20. PMID 36808186
- [Result] Conradie F, Bagdasaryan TR, Borisov S, Howell P, Mikiashvili L, Ngubane N, Samoilova A, Skornykova S, Tudor E, Variava E, Yablonskiy P, Everitt D, Wills GH, Sun E, Olugbosi M, Egizi E, Li M, Holsta A, Timm J, Bateson A, Crook AM, Fabiane SM, Hunt R, McHugh TD, Tweed CD, Foraida S, Mendel CM, Spigelman M; ZeNix Trial Team. Bedaquiline-Pretomanid-Linezolid Regimens for Drug-Resistant Tuberculosis. N Engl J Med. 2022 Sep 1;387(9):810-823. doi: 10.1056/NEJMoa2119430. PMID 36053506
- [Result] Nyang'wa BT, Berry C, Kazounis E, Motta I, Parpieva N, Tigay Z, Solodovnikova V, Liverko I, Moodliar R, Dodd M, Ngubane N, Rassool M, McHugh TD, Spigelman M, Moore DAJ, Ritmeijer K, du Cros P, Fielding K; TB-PRACTECAL Study Collaborators. A 24-Week, All-Oral Regimen for Rifampin-Resistant Tuberculosis. N Engl J Med. 2022 Dec 22;387(25):2331-2343. doi: 10.1056/NEJMoa2117166. PMID 36546625
- [Result] Nyang'wa BT, Berry C, Kazounis E, Motta I, Parpieva N, Tigay Z, Moodliar R, Dodd M, Solodovnikova V, Liverko I, Rajaram S, Rassool M, McHugh T, Spigelman M, Moore DA, Ritmeijer K, du Cros P, Fielding K; TB-PRACTECAL team. Short oral regimens for pulmonary rifampicin-resistant tuberculosis (TB-PRACTECAL): an open-label, randomised, controlled, phase 2B-3, multi-arm, multicentre, non-inferiority trial. Lancet Respir Med. 2024 Feb;12(2):117-128. doi: 10.1016/S2213-2600(23)00389-2. Epub 2023 Nov 16. PMID 37980911
- [Result] Zhang Y, Shi W, Zhang W, Mitchison D. Mechanisms of Pyrazinamide Action and Resistance. Microbiol Spectr. 2014 Aug;2(4):MGM2-0023-2013. doi: 10.1128/microbiolspec.MGM2-0023-2013. PMID 26104205
- [Result] Zhang Y, Chiu Chang K, Leung CC, Wai Yew W, Gicquel B, Fallows D, Kaplan G, Chaisson RE, Zhang W. 'Z(S)-MDR-TB' versus 'Z(R)-MDR-TB': improving treatment of MDR-TB by identifying pyrazinamide susceptibility. Emerg Microbes Infect. 2012 Jul;1(7):e5. doi: 10.1038/emi.2012.18. Epub 2012 Jul 25. PMID 26038418
- [Result] Fu L, Zhang X, Xiong J, Sun F, Weng T, Li Y, Zhang P, Li H, Yang Q, Cai Y, Liang H, Chen Q, Wang Z, Liu L, Chen X, Zhang W, Deng G. Selecting an appropriate all-oral short-course regimen for patients with multidrug-resistant or pre-extensive drug-resistant tuberculosis in China: A multicenter prospective cohort study. Int J Infect Dis. 2023 Oct;135:101-108. doi: 10.1016/j.ijid.2023.08.001. Epub 2023 Aug 10. PMID 37567554